CLINICAL TRIAL: NCT00266942
Title: The Determination of Differences Between Intr-Atrial vs. Extra-Cardiac Technique During the Fontan Operation: A Retrospective Review
Brief Title: Intra-Atrial vs. Extra-Cardiac Technique During Fontan Operation
Status: Terminated | Type: Observational
Why Stopped: data collection ended
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-109
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2007-05-23 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: Fontan procedure; single ventricle physiology; intra-atrial; extracardiac technique
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Our aim is a retrospective chart review seeking to determine any differences in the main clinical and outcome variables as well as general outcome data such as functional recovery, readmission rates, somatic growth and mortality. An n size of 150 to 200 for each of the 2 groups will give us excellent power to detect potential differences.

DETAILED DESCRIPTION:
The Fontan procedure is indicated as final-stage treatment for pediatric cardiac patients with single ventricle physiology. This procedure, whose aim is to provide for total cavopulmonary disconnect and perfusion of the pulmonary arteries via systemic veins, is performed via two differing techniques: intra-atrial, so-called lateral tunnel technique, employing PTFE graft material and internal atrial baffle, versus the extracardiac technique, using larger PTFE tubing and externally constructed baffle.

There is persistent debate regarding the optimal technique to use, centered around the following main issues: 1) need for use of cardiopulmonary bypass and attendant consequences, 2) rates of thrombosis and embolism, 3) incidence of postoperative protein-losing enteropathy (PLE), 4) incidence of arrhythmias, and 5) baffle patency rates. A handful of small- to medium-sized studies has addressed the above issues, but, importantly, has not used patient data from the same institution. Here at CHOA, there are an estimated 200+ lateral tunnel, and have been up to 125 to 150 extracardiac Fontan procedures, performed in the last 15 years (1.1.1980-3.31.2005). Data from these cases would be potentially very helpful in answering all of these questions.

ELIGIBILITY:
Inclusion Criteria:

* Children's Healthcare of Atlanta patients
* lateral tunnel procedure during 1.1.1990-3.31.2005
* extracardiac Fontan procedures during 1.1.1990 - 3.31.2005

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400
Dates: Start 1990-01; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Jason M. Budde, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States